CLINICAL TRIAL: NCT06271798
Title: Effect Of Resistive Exercises Versus Aerobic Exercises On Varicose Veins In Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Saif Elnasr Ghietah Hussein, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004867
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Varicose Veins
Keywords: Resistive Exercises; Aerobic Exercises; Varicose Veins; Postmenopausal Women
MeSH Terms: conditions — Varicose Veins | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Resistive exercise group): (Experimental): They will receive life style modification advice, in addition to performing resistive exercise three times per week for six weeks.
  Interventions: Other: Life style modification advice; Other: Resistive exercise
- Group B (Aerobic exercise group): (Experimental): They will receive the same life style modification advice, in addition to performing aerobic exercise three times per week for six weeks.
  Interventions: Other: Life style modification advice; Other: Aerobic exercises

INTERVENTIONS:
Other: Life style modification advice — The lifestyle modification advice involves several key elements: reducing daily standing periods, avoiding excessive flexion of the knee joint during sitting, weight reduction, addressing cardio-respiratory conditions, incorporating venotonic agents, and utilizing below-knee elastic compression devices. These measures collectively aim to mitigate the development and progression of varicose veins, potentially preventing complications such as deep venous thrombosis and improving overall circulatory health.
Other: Resistive exercise — Participants in group A will perform resistive exercise. The patients will be instructed to do seated toe raises exercise or standing toe raise exercise. The exercise will be performed for 30 minutes, three times per week for six weeks.
  Arms: Group A (Resistive exercise group):
Other: Aerobic exercises — Participants in group B will perform aerobic exercise. Each session will begin with 10 min of low-intensity treadmill walking for a warm-up. The subsequent aerobic component will involve incline treadmill walking for 20 min at a perceived exertion of 6-7 (i.e., somewhat hard) on Borg's 3-10 scale followed by 10 min of low-intensity treadmill walking for cool down. The exercise will be performed for 30 minutes, three times per week for six weeks.
  Arms: Group B (Aerobic exercise group):

SUMMARY:
The purpose of this study will be to determine the effect of resistive exercises on varicose veins in postmenopausal women, the effect of aerobic exercise on varicose veins in postmenopausal women and to compare between the effect of resistive exercise versus aerobic exercise on varicose veins in post menopausal women.

DETAILED DESCRIPTION:
Varicose veins in the lower extremities present a spectrum of symptoms from cosmetic issues to severe discomfort including telangiectases, reticular veins, edema, pigmentation, and venous ulceration. These veins lead to painful swelling, skin discoloration, and potential complications like thrombosis, and nerve injury, impacting an individual's efficiency and life quality. Exercise, particularly aerobic and resistance training, has shown promise in improving pain severity, functional ability, and venous blood flow.

So, the current study will be conducted to compare between the effect of resistive exercises versus aerobic exercises on varicose veins in postmenopausal women.

ELIGIBILITY:
Inclusion criteria:

* All women suffering from varicose veins.
* Their age will range from 50 to 65 years.
* Their body mass index will range from 25 to 29.9 kg/m2.
* Voluntary acceptance of participation in the study.

Exclusion Criteria:

* Had history of serious vascular disease as deep venous thrombosis.
* Sensory deficient
* Any dermatological condition that interferes with the procedure.
* Any musculoskeletal or neurological disorders.
* Acute or healed ulcer wounds.
* Any heart disease or pulmonary disease.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 44 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Peak popliteal vein velocity | 6 weeks
  It will be assessed by Doppler ultrasound scan for each woman in both groups before and after treatment.

SECONDARY OUTCOMES:
Visual analogue scale | 6 weeks
  It will be used to assess the leg pain intensity for each woman in both groups before and after treatment. The visual analogue scale is a 10 cm line with anchor statements on the left (no pain) and on the right (extra pain). Patients will be asked to mark their current pain level on the line.Then, the centimeters will be measured from the left end of the line to the marked point to obtain the score of leg pain intensity.
Chronic Venous Disease Quality of Life Questionnaire (CIVIQ-20) | 6 weeks
  It will be used to assess the quality of life for each woman in both groups before and after treatment. Patients will complete the self- questionnaire CIVIQ-20 in the waiting room. The secretary will hand out the questionnaire and collect it once completed. No particular assistance will be provided to patients. This procedure will be chosen on purpose to avoid any interference from an investigator. At study times, symptom severity will be quantified using a four-point scale (0 = absent, 1 = mild, 2 = significant, 3 = severe) for sensation of swelling, cramps and leg heaviness. The scores of CIVIQ-20 range from 0, the worst score, to 100, the best score.
6-minute. walk test | 6 weeks
  It is a sub-maximal test that will be used to assess the aerobic capacity and daily living activity for each woman in both groups before and after treatment procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Soheir Mahmoud Elkosery, PhD, Study Chair — Department of Woman's Health, Faculty of physical therapy, Cairo University, Giza, Egypt.
Locations (1):
- Cairo University, Giza, Egypt